CLINICAL TRIAL: NCT01554150
Title: A Randomised Controlled Trial Comparing Method of Levels Cognitive Therapy With a Contact Service for Improving Outcomes in Primary Care
Brief Title: Randomised Controlled Trial of Method of Levels Cognitive Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Timothy Bird, PhD Candidate, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11/NW/0736
Record Dates: First submitted 2012-03-12; First posted 2012-03-14 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-07

CONDITIONS: Mental Health Wellness 1; Depression; Anxiety
Keywords: Primary Health Care; Mental Health; Cognitive Therapy
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Method of Levels Cognitive Therapy (MOL) (Experimental): Participants in this arm will be able to receive therapy over a 3 month period. They will be able to schedule sessions with a therapist as and when they need them.
  Interventions: Behavioral: Method of Levels Cognitive Therapy
- Contact Service (No Intervention): The Contact Service arm is effectively a waiting list control. Participants assigned this arm will remain on the service's waiting list during the 3 months of the therapy phase. These participants will have access to a 'Contact Service' provided by the study therapist, where they are able to contact him if they want further information about the study or their treatment options.

INTERVENTIONS:
Behavioral: Method of Levels Cognitive Therapy — In MOL the therapist has two goals: to get the client to talk about his or her problem as it is currently being experienced, and to ask about disruptions, which are thought to indicate background thoughts coming into awareness. The assumption is that when somebody is experiencing problems that they feel they cannot solve, the only way for these to be properly resolved is for change to come from within that person. The MOL therapist helps the person redirect their awareness to think about the problem in more productive ways. It is present-focused, with the therapist asking questions relating to process rather than content. The therapist does not give advice and there is no homework. In MOL clients schedule sessions as and when they feel they need them and decide how long each session should be.
  Other Names: MOL
  Arms: Method of Levels Cognitive Therapy (MOL)

SUMMARY:
The purpose of this study is to determine whether Method of Levels Cognitive Therapy is an effective intervention for treating clients with a range of presenting problems in primary care by comparing it with a waiting list control condition.

ELIGIBILITY:
Inclusion Criteria:

* Anyone presenting to primary care services with mild to moderate mental health problems with capacity to provide informed consent and does not meet exclusion criteria.

Exclusion Criteria:

* Has been accepted into secondary care services.
* Aged under 16 years.
* Have an organic basis for their mental health problems. That is, mental health problems that are primarily caused by an identifiable brain malfunction such as thyroid problems or brain injury.
* Unable to provide informed consent.
* Is not able to speak, read, write or understand written and verbal English.
* Individuals who will be unable to understand and/or answer therapist questions due to learning disabilities, brain injury or similar neurological difficulties.
* Cannot attend sessions at the appropriate clinic.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire mood subscale (PHQ-9) | up to 3 months
Generalised Anxiety Disorder Assessment (GAD-7) | up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Warren Mansell, Principal Investigator — University of Manchester; Sara Tai, Principal Investigator — University of Manchester
Locations (1):
- Trafford Primary Care IAPT Services, Manchester, United Kingdom